CLINICAL TRIAL: NCT03498118
Title: Transversus Abdominis Plane Block Versus Wound Infiltration for Analgesia After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane Block Versus Wound Infiltration for Analgesia After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: aswu/200/2/18
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cesarean Section
Keywords: Transversus Abdominis Plane Block; Cesarean Delivery

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: the participants will be blinded to the medication type, which will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Abdominis Plane Block group (Experimental): after completion of surgery, 20 mL of bupivacaine 0.25% was injected under direct visualization in the plane between the transversus abdominis muscle and the fascia deep to the internal oblique muscle on each side.
  Interventions: Drug: 20 mL of bupivacaine 0.25%
- Wound Infiltration group (Active Comparator): at the end of surgery, 30 mL of bupivacaine 0.25% was injected subcutaneously into the surgical wound (15 mL in each of the upper and lower sides) by the obstetrician before skin closure
  Interventions: Drug: 20 mL of bupivacaine 0.25%

INTERVENTIONS:
Drug: 20 mL of bupivacaine 0.25% — In the infiltration group, at the end of surgery, 30 mL of bupivacaine 0.25% was injected subcutaneously in the surgical wound (15 mL in each of the upper and lower sides) by the obstetrician before skin closure. Sam procedure was performed by the primary investigator after completion of surgery by pressing a covered spinal needle on both sides of the patient's abdomen.
  In the TAP group, after completion of surgery, 20 mL of bupivacaine 0.25% was injected under direct visualization in the plane between the transversus abdominis muscle and the fascia deep to the internal oblique muscle on each side.
  Other Names: 30 mL of bupivacaine 0.25%

SUMMARY:
Adequate pain control after cesarean delivery is a major concern both for parturient and for obstetric anesthesiologists, and it usually comprises a combination of systemic and regional techniques.The transversus abdominis plane (TAP) block, affecting the nerves supplying the anterior abdominal wall, is a recently introduced, promising regional analgesic technique for a variety of abdominal and pelvic surgeries including cesarean delivery.(2,3) Infiltration of local anesthetic into the surgical wound (either as a single shot or using indwelling catheters) has long been used for postoperative analgesia.

Both the TAP block (4-6) and wound infiltration is superior to placebo; however, it is unknown which of them provides better analgesia after cesarean delivery because of a scarcity of randomized clinical trials. Only 2 studies compared the TAP block with wound infiltration after cesarean delivery with conflicting results, and another study compared it with continuous wound infusion and was prematurely terminated.

This study aimed to compare bilateral TAP block with single-shot local anesthetic wound infiltration for analgesia after cesarean delivery performed under spinal anesthesia. We hypothesized that the TAP block would decrease postoperative cumulative opioid consumption at 24 hours

DETAILED DESCRIPTION:
The study will conduct at the obstetric department of ASWAN University Hospital in ASWAN, Egypt, from January 2018 to the end of January 2019. Eligible subjects were American Society of Anesthesiologists physical status I, II parturient with full-term singleton pregnancies undergoing elective cesarean delivery under spinal anesthesia.

Exclusion criteria were: <19 years of age or >40 years of age; height <150 cm, weight <60 kg, body mass index (BMI) >=40 kg/m2; contraindications to spinal anesthesia (increased intracranial pressure, coagulopathy, or local skin infection); history of recent opioid exposure; hypersensitivity to any of the drugs used in the study; significant cardiovascular, renal, or hepatic disease; and known fetal abnormalities.

The study subjects will randomly have assigned to 2 equal groups (infiltration and TAP groups) using a computer-generated table of random numbers. A single investigator assessed the patients for eligibility, obtained written informed consent, and recorded the baseline data for each participant during the preanesthetic interview on the day of delivery. Sequentially numbered, sealed opaque envelopes containing group allocation were opened by the primary investigator after administration of spinal anesthesia. Neither the study subjects nor the outcome assessors knew the study group. The patients were separated from the surgical field and the operators by a large opaque screen. The primary investigator, who had experience in TAP block, performed the TAP block and the Sam procedure after closure of the skin when the patients were still lying on the operating table. The local anesthetic wound infiltration was performed by the operating obstetrician. An obestetrician resident who was not involved in the study, will record the intraoperative data and prepare, as instructed by the primary investigator, the local anesthetic solution for the TAP block and wound infiltration. The outcome data (opioid consumption, , pain scores, level of sedation, side effects, and patient satisfaction) were recorded by a blinded investigator who visited the patient in the ward at 2, 4, 6, 12, and 24 hours postoperatively.

No premedication was administered. Standard monitors (noninvasive blood pressure, electrocardiography, and pulse oximetry) were applied, and spinal anesthesia was administered in the sitting position at the L3-L4 or L4-L5 interspace using a 27-gauge or 25-gauge spinal needle; 12.5 mg of hyperbaric bupivacaine (2.5 mL 0.5%) and 15 µg of fentanyl were intrathecally administered. Surgery started after attaining an upper sensory level of T6 or higher, tested with pinprick. If the upper sensory level was below T6 after 20 minutes, this was considered a failed spinal, and the patient would have been excluded from the study. Lower segment cesarean delivery was performed using the Pfannenstiel incision, and exteriorization of the uterus was done in all cases. The upper sensory level was assessed using pinprick 30 minutes after intrathecal injection and recorded. If the patient complained of abdominal pain or discomfort after the start of surgery, 2 mg of intravenous (IV) midazolam was administered. If pain or discomfort persisted after midazolam administration, IV fentanyl and Propofol were administered as appropriate, and the patient was excluded from the study.

In the infiltration group, at the end of surgery, 30 mL of bupivacaine 0.25% was injected subcutaneously in the surgical wound (15 mL in each of the upper and lower sides) by the obstetrician before skin closure. Sam procedure was performed by the primary investigator after completion of surgery by pressing a covered spinal needle on both sides of the patient's abdomen.

In the TAP group, after completion of surgery, 20 mL of bupivacaine 0.25% was injected under direct visualization in the plane between the transversus abdominis muscle and the fascia deep to the internal oblique muscle on each side.

Duration of surgery (time from the start of skin incision to the end of skin closure) was recorded.The study subjects received postoperative standard analgesia according to their pain scale At 2, 4, 6, 12, and 24 hours postoperatively, the severity of pain at rest and on movement (hip flexion and coughing) was assessed using an 11-point numerical rating scale (0 = no pain and 10 = the worst possible pain). Patient satisfaction from postoperative analgesia was assessed at 24 hours postoperatively using a 5-point scale (1 = very unsatisfied, 2 = unsatisfied, 3 = fair, 4 = satisfied, and 5 = very satisfied(.

The primary outcome was cumulative opiod consumption at 24 hours. Secondary outcomes were the time to the first postoperative fentanyl dose, cumulative fentanyl consumption at 2, 4, 6, and 12 hours, pain scores at rest and on movement at 2, 4, 6, 12, and 24 hours, the deepest level of sedation, the incidence of side effects (nausea and vomiting and pruritis), and patient satisfaction.

Statistically analysis:

Data were entered and statistically analyzed using the Statistical Package for Social Sciences (SPSS) version 16. Qualitative data were described as numbers and percentages. Chi-square test and Monte Carlo test were used for comparison between groups, as appropriate. Quantitative data were described as means (SD) or medians, as appropriate. They were tested for normality by Kolmogorov-Smirnov test. In the normally distributed variables, one-way ANOVA test with LSD post-hoc multiple comparisons was used for comparison between groups. In the non-normally distributed variables, Kruskal-Wallis test was used for comparison between groups. -Odds ratios and their 95% confidence interval were calculated. "p-value ≤0.05" was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were American Society of Anesthesiologists physical status I, II parturient with full-term singleton pregnancies undergoing elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* were: <19 years of age or >40 years of age; height <150 cm, weight <60 kg, body mass index (BMI) >=40 kg/m2; contraindications to spinal anesthesia (increased intracranial pressure, coagulopathy, or local skin infection); history of recent opioid exposure; hypersensitivity to any of the drugs used in the study; significant cardiovascular, renal, or hepatic disease; and known fetal abnormalities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
pain score after cesarean section in the first 24 hour posoperative | 24 hours post operaive
  pain score after cesarean section in the first 24 hour posoperative

SECONDARY OUTCOMES:
cumulative opioid consumption at 24 hours | 24 hours post operaive
  cumulative opioid consumption at 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- AswanUH, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No